CLINICAL TRIAL: NCT03906084
Title: Evaluation of the Combined Effect of Corticotomy and Low Level Laser Therapy on the Rate of Orthodontic Tooth Movement: Split Mouth Randomized Clinical Trial
Brief Title: Evaluation of the Effect of Corticotomy and Low Level Laser Therapy on Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Ahmed Farid Shehab, Assistant lecturer, Orthodontics department, Faculty of Dentistry-MSA University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2015-03-17
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Dental Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind Endpoint Classification: Efficacy Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticotomy facilitated orthodontics. (Active Comparator): Corticotomy is carried out under local anesthesia in right side.
  Interventions: Procedure: Corticotomy and low laser therapy
- Corticotomy and low level laser therapy (Experimental): Corticotomy is carried out under local anesthesia followed by low-intensity laser therapy that is started on the selected experimental side on the same day as placement of the coil spring
  Interventions: Procedure: Corticotomy facilitated Orthodontics

INTERVENTIONS:
Procedure: Corticotomy and low laser therapy — Corticotomy is carried out under local anesthesia followed by low-intensity laser therapy that is started on the selected experimental side on the same day as placement of the coil spring
  Arms: Corticotomy facilitated orthodontics.
Procedure: Corticotomy facilitated Orthodontics — Corticotomy is carried out under local anesthesia in right side.
  Arms: Corticotomy and low level laser therapy

SUMMARY:
The aim of the present study was to compare, a standard efficient technique in accelerating OTM as surgical corticotomy as a gold standard versus surgical corticotomy combined with LLLT in an attempt for further acceleration of OTM.

DETAILED DESCRIPTION:
The study design was a randomized split mouth design to compare, clinically and radiographically, between the two interventions (Corticotomy and Laser versus Corticotomy only) by assessing the rate of maxillary canine retraction achieved in 4 months. Secondary outcomes were to evaluate 1st maxillary molar anchorage loss, changes in tipping, torque and rotations values of maxillary canine and 1st molar. In addition, the impact of both interventions on root resorption was assessed. The present study was carried on 16 female patients. All patients required maxillary 1st premolar extraction and subsequent maxillary canine retraction.

ELIGIBILITY:
Inclusion Criteria:

1. Post pubertal patients with age more than 17 years.
2. Class I or Class II (Angles' classification) malocclusion cases requiring 1st premolar extraction with moderate anchorage.

Exclusion Criteria:

1. Patients having missing permanent canine teeth in maxillary arch.
2. History of trauma or root canal treatment in maxillary canines.
3. History of previous orthodontic treatment.
4. History of hormonal disorder or syndrome.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction | 4 months
  Rate of canine retraction using a digital caliper, units of mm, readings extracted from digital models reading each month.

SECONDARY OUTCOMES:
Root resorption | after 4 months from start of clinical trial
  Root resorption using CBCT in mm after the end of canine retraction period (at the end of 4 months)